CLINICAL TRIAL: NCT00495222
Title: Evaluation of an Endoscopic Suturing System for Tissue Apposition
Brief Title: Endoscopic Suturing System for Tissue Apposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Susan Knippenberg, Ethicon Endo-Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-06-0005
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Obesity
Keywords: gastrojejunostomy; stoma
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tissue plication (Experimental): The Endoscopic Suturing System (ESS) is used for tissue apposition and reduction of the size of a dilated GJ anastomosis in subjects who are regaining weight after successful weight loss following gastric bypass
  Interventions: Procedure: Tissue plication; Device: Endoscopic Suturing System; Device: Tissue Plication

INTERVENTIONS:
Procedure: Tissue plication — Tissue apposition and plication of a dilated GJ anastomosis with the Endoscopic Suturing System
Device: Endoscopic Suturing System — Tissue plication of dilated GJ stoma
Device: Tissue Plication — Tissue plication for GJ stoma reduction

SUMMARY:
The objective of this feasibility trial is to evaluate the Ethicon Endo-Surgery Endoscopic Suturing System (ESS) for tissue apposition and reduction of the size of a dilated GJ anastomosis in subjects who are regaining weight after successful weight loss following gastric bypass. Post-procedure weight will be followed to assess whether weight loss is resumed.

The ESS is an FDA-cleared (510(k)) sterile, single-use, disposable suturing system indicated for endoscopic placement of suture(s) and approximation of soft tissues. It is designed to facilitate endoscopic gastrointestinal procedures.

ELIGIBILITY:
Inclusion Criteria

Subjects must fulfill the following criteria to be entered in this study:

* Review and sign informed consent;
* Between 21 and 65 years of age (inclusive) at time of trial enrollment;
* Documented Roux-en-Y Gastric Bypass (RYGB) surgery date
* Documented baseline weight at the time of RYGB procedure;
* > 12 months post RYGB);
* Body mass Index (BMI) > 30 and at least 20 pounds in excess of post-RYGB weight nadir;
* Patients initially achieved at least 50% excess weight loss (EWL) post RYGB;
* Visible anastomotic junction (between gastric pouch and the Roux-limb);
* Stoma size at screening > 15mm; and
* Negative serum pregnancy test for women of childbearing potential.

Exclusion Criteria

Subjects will be excluded from the trial for any of the following:

* Documented history of esophageal pathology (e.g., esophageal varices, Barrett's Esophagus);
* American Anesthesia Association (ASA) Class IV or V and/or any contraindications to monitored anesthesia;
* Documented history of GJ anastomosis stricture (within 6 months);
* Documented history of previous RYGB revision;
* Presence or documented presence of gastric/duodenal ulcers;
* Presence of sepsis;
* Medical or physical endoscopic contraindications, including esophageal varices or bleeding, laryngeal perforation, trauma to pharynx, aspiration pneumonia, acute peritonitis, and other conditions where general endoscopic techniques and/or placement of overtube are contraindicated;
* Chronic Non-Steroidal Anti-Inflammatory Drug (NSAID) use (subjects taking a single aspirin tablet per day for cardioprotection are considered acceptable);
* Uncontrolled diabetes;
* Physical or psychological condition which would impair trial participation per investigator discretion;
* Binge-eating or similar eating disorders;
* Unable or unwilling to attend follow-up visits and examinations;
* Concurrent surgical procedure (intra-operative exclusion during ESS procedure);
* Participation in any other investigational device or drug trial within 30 days prior to enrollment; or
* Any condition, which precludes compliance with the trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Torquati, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tissue Plication
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tissue Plication
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Knotting Elements Placed
Description: completion of plication (1-3 knotting elements placed per procedure)
Time Frame: intra-operative
Population: Intent to Treat
Measure: Number; unit: elements
Arm/Group | Tissue Plication
Number analyzed (Participants) | 9
elements | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No